CLINICAL TRIAL: NCT04982133
Title: Randomised Trial Weight Gain in Extremely Premature Infant: Targeted Versus Adjusted Fortification
Brief Title: Weight Gain in Extremely Premature Infant With Targeted Versus Adjusted Fortification
Acronym: FORTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Esperanza Escribano, Co-investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HULP5704
Record Dates: First submitted 2021-07-05; First posted 2021-07-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Preterm; Very Low Birth Weight Infant; Feeding, Breast; Food, Fortified
Keywords: preterm; nutrition; human milk fortified
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortification adjusted according to urea (Active Comparator): Fortification adjusted according to urea with FM 85 at 4% and oligopeptides. In this arm, fortification at 4% is started, and according to plasma urea control every 15 days the fortification is modified.
  Interventions: Dietary Supplement: Protein supplementation based on plasma urea concentration every other week or human milk analysis on experiment
- Individualized fortification according to the nutritional characteristics of breast milk (Experimental): Individualized fortification according to the nutritional characteristics of the mother's own milk or pasteurized milk taken by the premature infant.
  In this arm, fortification is adjusted based on the macronutrient analysis of breast milk or donated twice weekly.
  Interventions: Dietary Supplement: Protein supplementation based on plasma urea concentration every other week or human milk analysis on experiment

INTERVENTIONS:
Dietary Supplement: Protein supplementation based on plasma urea concentration every other week or human milk analysis on experiment — At the time that the doctor decides to start fortification, it will be done according to urea levels in active comparator arm or human milk analysis on experimental group.
  In Group A, fortification at 4% is started, and according to plasma urea control every 15 days the fortification is modified.
  In Group B, fortification is adjusted based on the macronutrient analysis of breast or donated milk.
  Other Names: Macronutrient supplementation based on human milk analysis

SUMMARY:
Investigation about the effect on weight gain in extremely low birth weight preterm with individualized fortification, according to human milk analysis versus fortification adjusted according to urea serum concentration.

DETAILED DESCRIPTION:
1. Study design This is an interventional, randomized, controlled study.
2. Description of the study The very premature newborn will be identified by daily evaluation of the infants admitted for consultation in the income book.

   Informed consent will be requested from the infant´s father, mother or legal guardian between the fifth and tenth day of life.

   Fortification will be done according to the randomization group.
3. Outline of the study design

   * Excel calculation sheet of individualized supplementation according to the composition of breast milk in the target fortification group. Methodology of analysis of breast milk in FOSS analyzer.
   * In the adjusted fortification group, urea concentration levels will be kept between 19-30 mg / dL
   * Fenton curves or https://www.growthcalculator.org/ will be used for Z-scores calculation.
   * Growth speed calculation: Weight gain: (1000x ln [Final weight / Initial weight]) / number of days.

     4 Duration of the study for each participant The duration of participation in the study and the fortification intervention period will be a maximum of 132 days.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born <1000 g of birth weight that are fed with breast milk or donated milk.
2. Written informed consent signed by the mother, father or legal guardian.
3. To tolerate enteral feeding, at least 100mL / kg / day.

Exclusion Criteria:

1. Non-premature or premature patients weighing ≥ 1000 gr.
2. Patients with major malformations.
3. Patients with diagnosed chromosomal diseases or of high diagnostic suspicion.
4. Patients with short bowel syndrome or any surgery on the gastrointestinal tract.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Growth rate 28 days after the start of fortification and birth | 28 days
  To investigate the effect on weight gain during admission of individualized fortification, according to milk analysis, versus fortification adjusted according to urea level.

SECONDARY OUTCOMES:
Mineralization differences between both fortication methods | Until 36 weeks of postmenstrual age (EPM) or at discharge
  Difference in phosphate and alkaline phosphatase values

CONTACTS AND LOCATIONS:
Overall Officials: MARTA CABRERA, Principal Investigator — La Paz University Hospital
Locations (1):
- University Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the results reported in this article after deidentification (text, tables, figures and appendices) will be available upon request. Data will be available 3 months to 5 years after publication of the article. Other documents will be available: study protocol, informed consent form. Researchers submitting a methodologically sound proposal should contact miguel.saenz@salud.madrid.org. In order to access, requesters will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 3 months to 5 years after publication of the article.
Access Criteria: Researchers submitting a methodologically sound proposal should contact miguel.saenz@salud.madrid.org. In order to access, requesters will need to sign a data access agreement.